CLINICAL TRIAL: NCT06602843
Title: Neoadjuvant Chemoimmunotherapy Followed by Surgery and Postoperative Radioimmunotherapy in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Chemoimmunotherapy Followed by Surgery and Postoperative Radioimmunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-042
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Locally advanced; Chemoimmunotherapy; Radioimmunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Neoadjuvant chemoimmunotherapy followed by surgery and postoperative radioimmunotherapy
  Interventions: Procedure: Neoadjuvant chemoimmunotherapy followed by surgery and postoperative radioimmunotherapy
- Comparator (Active Comparator): chemoradiotherapy followed by surgery
  Interventions: Procedure: Neoadjuvant chemoimmunotherapy followed by surgery and postoperative radioimmunotherapy

INTERVENTIONS:
Procedure: Neoadjuvant chemoimmunotherapy followed by surgery and postoperative radioimmunotherapy — Neoadjuvant chemoimmunotherapy followed by surgery and postoperative radioimmunotherapy

SUMMARY:
The goal of this study was to explore the efficacy and safety of neoadjuvant chemoimmunotherapy followed by surgery and postoperative radioimmunotherapy in patients with locally advanced esophageal squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75;
* Radical operation for esophageal cancer;
* Esophageal squamous cell carcinoma was confirmed by postoperative pathology; . Preoperative imaging (enhanced cervical, thoracoabdominal CT+ bone scan) and postoperative pathological evaluation were performed, and the stage was pIIB-IVA (AJCC eighth edition staging criteria: T≥3 or N+).
* More than or equal to 12 lymph nodes were surgically removed;
* Postoperative ECOG score 0-1, able to tolerate postoperative adjuvant radiotherapy and immunotherapy;
* Informed consent signed by patient or family member.

Exclusion Criteria:

* Less than 18 years old, more than 75 years old;
* did not receive radical resection of esophageal cancer, including palliative resection;
* Postoperative pathology showed non-esophageal squamous cell carcinoma;
* After preoperative imaging (enhanced cervical, thoracoabdominal CT+ bone scan) and postoperative pathological evaluation, the stage was pI, IIA, IVB (AJCC eighth edition staging standard); e. Less than 12 lymph nodes were surgically removed;
* Postoperative ECOG score 2-3 points, unable to tolerate postoperative adjuvant radiotherapy and immunotherapy;
* The patient or family member did not sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | immediately after the intervention/procedure/surgery
  Pathologic Complete Response

SECONDARY OUTCOMES:
R0 resection rate | immediately after the intervention/procedure/surgery
  R0 resection rate

OTHER OUTCOMES:
1#3-year disease free survival | immediately after the intervention/procedure/surgery
  1#3-year disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui provincial hospital, Hefei, China

IPD SHARING:
Plan to Share IPD: Undecided